CLINICAL TRIAL: NCT00945256
Title: A Phase I Trial Examining Muscle Perfusion and Protein Metabolism in Elderly and Young
Brief Title: Muscle Perfusion and Protein Metabolism in Elderly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: 03-213; R01AG021539 (NIH)
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Results first posted 2016-01-05 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2014-04

CONDITIONS: Aging
Keywords: metabolism; exercise; sodium nitroprusside
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Nitroprusside

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Young Aerobic Exercise (Active Comparator): 45 minutes of treadmill walking at 40% VO2 peak
  Interventions: Other: Aerobic Exercise
- Elderly Aerobic Exercise (Active Comparator): 45 minutes of treadmill walking at 40% VO2 peak
  Interventions: Other: Aerobic Exercise
- Young Sodium Nitroprusside (Active Comparator): Sodium Nitroprusside given in a constant infusion for 180 minutes at a rate of 0.114 ug/kg/min
  Interventions: Drug: Sodium Nitroprusside
- Elderly Sodium Nitoprusside (Active Comparator): Sodium Nitroprusside given in a constant infusion for 180 minutes at a rate of 0.114 ug/kg/min
  Interventions: Drug: Sodium Nitroprusside
- Elderly Sodium Nitroprusside and Amino Acid Drink (Active Comparator): Sodium Nitroprusside given in a constant infusion for 180 minutes at a rate of 0.114 ug/kg/min and 7.5g amino acid drink taken orally
  Interventions: Drug: Sodium Nitroprusside; Dietary Supplement: Amino Acid Drink

INTERVENTIONS:
Other: Aerobic Exercise — 45 minuties of treadmill walking was completed at 40% VO2 peak
  Arms: Elderly Aerobic Exercise; Young Aerobic Exercise
Drug: Sodium Nitroprusside — Sodium Nitroprusside was given in a constant infusion for 180 minutes at a rate of 0.114 ug/kg/min
  Other Names: Nitropress
  Arms: Elderly Sodium Nitoprusside; Elderly Sodium Nitroprusside and Amino Acid Drink; Young Sodium Nitroprusside
Dietary Supplement: Amino Acid Drink — 7.5 gram Amino Acid drink
  Arms: Elderly Sodium Nitroprusside and Amino Acid Drink

SUMMARY:
The purpose of this study was to examine the role skeletal muscle perfusion plays in mediating muscle protein synthesis in healthy older and younger individuals. The investigators hypothesized that normalization of muscle perfusion in older men and women via exercise or infusion of a vasodilator would enhance nutritive flow and skeletal muscle protein synthesis in the elderly similar to that of their younger counterparts.

DETAILED DESCRIPTION:
The purpose of this study was to examine muscle protein metabolism in healthy young and elderly subjects during pharmacologic vasodilation of the lower limb vasculature in combination with increased amino acids delivery. We obtained femoral arteriovenous blood samples and v. lateralis muscle biopsies during a primed continuous infusion of L-[ring-13C6] Phenylalanine. Muscle protein kinetics were measured in the basal state and during a 180 min infusion of sodium nitroprusside (SNP) and amino acids (Premsol 10%) (SNP+AA). Skeletal muscle microvascular recruitment and flow were measured during the basal state and SNP+AA using contrast-enhanced ultrasound (CEU).

ELIGIBILITY:
Inclusion Criteria:

All inclusion criteria must be fulfilled throughout the study. At enrollment, subjects must fit the following criteria:

1. Age: young 18-40 yrs; elderly 60-85 yrs.
2. Availability of transportation (i.e., subjects must be able to provide their own transportation to UTMB).
3. Ability to sign informed consent (score >24 on 30 item mini-mental status exam and no errors on assessment of judgment).

Exclusion Criteria:

None of the following exclusion criteria should be present at enrollment or throughout the study:

1. Patients with limiting or unstable angina or who demonstrate cardiac abnormalities such as > 0.2 mV horizontal or downsloping ST segment depression, frequent arrhythmias (>10 PVC/min), or valvular disease.
2. Any patient with atrial fibrillation, history of syncope, angina, or congestive heart failure.
3. Patients with vascular disease, as determined by the presence of risk factors of peripheral atherosclerosis (i.e., hypertension, obesity, uncontrolled diabetes, and evidence of venous or arterial insufficiency upon palpation of femoral, popliteal, and pedal arteries).
4. Peripheral vascular disease as determined by history or abnormal ankle-brachial index by Doppler (< 1.0).
5. Any subject with blood pressure on three consecutive measurements taken at rest on separate occasions that has a systolic pressure >170 mm Hg or a diastolic blood pressure >100 mm Hg will be excluded. Subjects will not be included if they are taking blood pressure medication and have a blood pressure above these criteria.
6. Any person HIV-seropositive, with active hepatitis, or any other immunosuppressive or autoimmune disease.
7. Any patient taking beta blockers, vasodilators, angiotensin-converting enzyme inhibitors, calcium channel blockers, or alpha blockers.
8. Any patient with uncontrolled metabolic diseases including any patient with liver or renal disease.
9. Glucose intolerance: fasting plasma glucose concentration 110-126 mg/dL (6.1-7 mmol/L) and/or 2-h plasma glucose 140-200 mg/dL (7.8-11.1 mmol/L) during oral glucose tolerance test (OGTT).
10. Currently in muscle strengthening program.
11. Total knee replacement or moderate to severe degenerative joint disease of knees.
12. Anemia (hemoglobin <13 g/dL in males or <12 g/dL in females).
13. Any history of hypo- or hyper-coagulation disorders, including patients taking Coumadin or with a history of deep venous thrombosis (DVT) or pulmonary embolism (PE) at any point in their lifetimes.
14. Currently taking aspirin and cannot stop for 7 days (i.e., medical indication for continued aspirin such as transient ischemic attacks).
15. Presence of acute illness or metabolically unstable chronic illness.
16. Heart disease requiring therapy or recent myocardial infarction (less than 1 year)
17. Currently on weight-loss diet.
18. Active cancer or in short-term remission (less than 3 years).
19. Alcohol or drug abuse.
20. History of >20 packs per year cigarette smoking.
21. Recent (within 6 months) ingestion or injection or transdermal administration of anabolic steroids, corticosteroids, estrogens, or progestagens.
22. History of falls (1 fall in the past year which required medical attention, or more than 2 falls/year regardless of severity).
23. Allergy to iodides, penicillin or shellfish.
24. Any subject with a know hypersensitivity to octafluoropropane.
25. Any subject with a cardiac shunt.
26. Any subject with chronic obstructive pulmonary disease (COPD).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2003-05; Primary Completion 2008-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Sheffield-Moore, PhD, Principal Investigator — UTMB

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Young groups: Ages 18 - 40; Elderly groups: Ages 60 - 85
Groups:
- Young Aerobic Exercise: 45 minutes of treadmill walking completed at 40% VO2 peak
- Young Sodium Nitroprusside; Elderly Sodium Nitroprusside: Sodium Nitroprusside (Nitropress) given in a constant infusion for 180 minutes at a rate of 0.114 ug/kg/min.
- Elderly Sodium Nitroprusside and Amino Acid Drink: Sodium Nitroprusside (Nitropress) given in a constant infusion for 180 minutes at a rate of 0.114 ug/kg/min and 7.5 gram amino acid drink taken orally.
Period: Overall Study
Arm/Group | Young Aerobic Exercise | Elderly Aerobic Exercise | Young Sodium Nitroprusside | Elderly Sodium Nitroprusside | Elderly Sodium Nitroprusside and Amino Acid Drink
Started | 13 | 10 | 15 | 16 | 8
Completed | 9 | 8 | 7 | 7 | 7
Not Completed | 4 | 2 | 8 | 9 | 1

BASELINE CHARACTERISTICS:
Groups:
- Elderly Aerobic Exercise: 45 minutes of treadmill walking completed at 40% VO2 peak.
- Total: Total of all reporting groups
Arm/Group | Young Aerobic Exercise | Elderly Aerobic Exercise | Young Sodium Nitroprusside | Elderly Sodium Nitroprusside | Elderly Sodium Nitroprusside and Amino Acid Drink | Total
Number analyzed (Participants) | 13 | 10 | 15 | 16 | 8 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 3 | 15 | 6 | 5 | 42
  >=65 years | 0 | 7 | 0 | 10 | 3 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (5.9) | 67.4 (5.1) | 26.4 (5.0) | 68.1 (5.9) | 67.1 (4.4) | 49.2 (21.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 10 | 7 | 7 | 24
  Male | 13 | 10 | 5 | 9 | 1 | 38
Region of Enrollment [Number; unit: participants]
  United States | 13 | 10 | 15 | 16 | 8 | 62

OUTCOME MEASURES:

1. Primary Outcome: Mixed Muscle Fractional Synthesis Rate (FSR)
Description: The rate at which the body makes new muscle was assessed by determining the fractional synthesis rate (FSR). This technique determines how quickly new amino acids are used to make muscle. In this technique, a special (but natural and non-radioactive) version of an amino acid is infused into the blood. This special version of the amino acid is heavier than the most common version the same amino acid. This property allows it to be identified in a muscle sample. By determining how much of the special amino acid has accumulated over time in a muscle sample, the fractional synthesis rate can be determined. For example, if the rate were such that 1 of every 100 amino acids were of the special type after 1 day, the fractional synthesis rate would be 1% per day. In other words, 1/100 of the muscle would be newly made each day.
Time Frame: Acute ( 8 hours)
Population: FSR was not calculated for the Elderly Sodium Nitroprusside with Amino Acid Drink arm of the study.
Measure: Mean (Standard Error); unit: Fractional Synthesis Rate (pecent/hour)
Groups:
- Elderly Sodium Nitroprusside (SNP): Sodium Nitroprusside (Nitropress) given in a constant infusion for 180 minutes at a rate of 0.114 ug/kg/min.
- Elderly Sodium Nitroprusside and Amino Acid Drink: Sodium Nitroprusside (Nitropress) given as a constant infusion for 180 minutes at a rate of 0.114 ug/kg/min and a 7.5g amino acid drink taken orally.
Arm/Group | Young Aerobic Exercise | Elderly Aerobic Exercise | Young Sodium Nitroprusside | Elderly Sodium Nitroprusside (SNP) | Elderly Sodium Nitroprusside and Amino Acid Drink
Number analyzed (Participants) | 13 | 10 | 15 | 16 | 8
Fractional Synthesis Rate (pecent/hour)
  Pre-intervention (either exercise or SNP) | 0.061 (0.005) | 0.070 (0.006) | 0.066 (0.01) | 0.070 (0.004) | NA (NA) — FSR was not calculated for this arm of the study.
  Post -intervention (either exercise or SNP) | 0.098 (0.009) | 0.111 (0.011) | 0.090 (0.008) | 0.095 (0.009) | NA (NA) — FSR was not calculated for this arm of the study.

ADVERSE EVENTS:
Time Frame: Time frame for Adverse Event Reporting is the study date and one week past the study date to assess any problems with muscle biopsies, catheter placement.
Description: Adverse events were self reported by subjects to clinical research staff.
Groups:
- Young Sodium Nitroprusside; Elderly Sodium Nitroprusside: Sodium Nitroprusside (Nitropress) given as a constant infusion for 180 minutes at a rate of 0.114 ug/kg/min.
- Elderly Sodium Nitroprusside and Amino Acid Drink: Sodium Nitroprusside (Nitropress) given as a constant infusion for 180 minutes at a rate of 0.114 ug/kg/min and 7.5 grams of amino acids taken orally.
Arm/Group | Young Aerobic Exercise | Elderly Aerobic Exercise | Young Sodium Nitroprusside | Elderly Sodium Nitroprusside | Elderly Sodium Nitroprusside and Amino Acid Drink
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/10 | 0/15 | 1/16 | 0/8
Other Adverse Events (participants affected / at risk) | 0/13 | 0/10 | 2/15 | 2/16 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Young Aerobic Exercise (N=13) | Elderly Aerobic Exercise (N=10) | Young Sodium Nitroprusside (N=15) | Elderly Sodium Nitroprusside (N=16) | Elderly Sodium Nitroprusside and Amino Acid Drink (N=8)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — The subject developed cellulitis near the placement of the femoral catheters 3 days post procedure.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Young Aerobic Exercise (N=13) | Elderly Aerobic Exercise (N=10) | Young Sodium Nitroprusside (N=15) | Elderly Sodium Nitroprusside (N=16) | Elderly Sodium Nitroprusside and Amino Acid Drink (N=8)
Redness at biopsy site (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Swelling at femoral catheter site (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Back pain in direct relation to infusion of Definity Microbubbles

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No